CLINICAL TRIAL: NCT02488200
Title: Peridialysis Project: The Influence of Predialysis Factors on the Initial Course of Dialysis
Acronym: Peridialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital Skejby (Other); Zealand University Hospital (Other); Holbaek Sygehus (Other); Central Jutland Regional Hospital (Other); Sonderborg Hospital (Other Government); Skovde Hospital (Unknown); Karolinska University Hospital (Other); Lund University Hospital (Other); Turku University Hospital (Other Government); Pauls Stradins Clinical University Hospital (Other); Tartu University Hospital (Other); The Hospital of Vestfold (Other); St. Olavs Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, James heaf, Doctor, Herlev Hospital
Other Study IDs: CRU ID 15002474
Record Dates: First submitted 2015-06-13; First posted 2015-07-02 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The present study plans to delineate the clinical, biochemical, sociological and psychological factors. involved in dialysis preparation, and their impact on dialysis initiation (DI), modality choice and prognosis. In particular the following questions are to be answered.

1. What factors influence unplanned DI?
2. What factors influence choice of dialysis modality?
3. What factors influence choice of dialysis access?
4. Why do physicians start dialysis?
5. What factors in the predialytic period and its immediate aftermath (the "peridialytic" period) influence prognosis?

DETAILED DESCRIPTION:
Patients All patients starting active end stage renal disease (ESRD) treatment at the participating centres and their satellite centres.

No. Patients: 1000.

1. Patients who have received their recent predialysis care at another centre can be included if the previous centre's notes are available, otherwise not.
2. Patients receiving a preemptive transplant are included, even if the transplant is performed at another centre. A patient questionnaire is not required for these patients.
3. Africans are excluded (inaccurate estimated glomerular filtration rate (eGFR) calculation) Each patient is allocated a local identity number (1,2,3….). The local author keeps a registry of the true patient identity of each identity number for follow-up purposes. This registry is not to be used in any communication outside the centre.

Comment: Most patients have known chronic uremia at dialysis start. In a few cases, it is unknown whether the uremia is acute or chronic. There are two main groups:

1. Acute uremia of unknown origin. Doctors should fill the questionnaire in Table 2, which can be discarded if the patient recovers renal function within three months.
2. Acute kidney injury (AKI). Most of these patients will recover within three months, so the questionnaire can wait, and be filled in retrospectively for the few remaining patients.

Methods

1. Each participating centre fills a Centre Questionnaire, see Table 1.
2. All prescribing doctors fill in a voluntary Physician Questionnaire, see Table 4.
3. The doctor prescribing the first dialysis fills in a Motivation Questionnaire, see Table 2.
4. The local coordinator fills in a Patient Notes Review

   1. Birthday
   2. Sex
   3. Height and weight
   4. Renal diagnosis
   5. Comorbidity
   6. Date and creatinine at referral to nephrology dept.
   7. Date and creatinine 6 months before dialysis start
   8. Date and creatinine 3 months before dialysis start
   9. Date and creatinine at start of dialysis information/choice
   10. Date and creatinine at access prescription. Date and creatinine at access creation. If there are several attempts at access creation, the last attempt is registered. For unplanned dialysis start, this is often the same date as dialysis start.
   11. Date of dialysis start
   12. Following values before first dialysis: B-hemoglobin, p- creatinine, urea, potassium, calcium, phosphate, bicarbonate, albumin
   13. Initial dialysis modality (centre hemodialysis (HD)/Home HD/continuous ambulatory peritoneal dialysis (CAPD)/ automated peritoneal dialysis (APD))
   14. Type of start (Planned/unplanned)
   15. Reason for unplanned start (primary and (if appropriate) secondary).
   16. For hemodialysis patient (HD) patients, initial access (areteriovenous fisula (AVF)/arteriovenous graft (AVG) /tunneled central venous catheter (CVC)/temporary CVC)
   17. Modality after 3 months (Center HD/Home HD/CAPD/APD/regained function/Transplanted/Dead)
   18. Is the patient alive after 3 months Yes/No. If "No" Date of death.
   19. Is the patient alive after 6 months Yes/No.
   20. If "No" Date of death.Is the patient alive after 12 months Yes/No. If "No" Date of death.
   21. Was the patient transplanted after inclusion? If so, when?

Responsibilities National coordinators are responsible for translation of protocol to local language, and compliance with any necessary national regulatory requirements (data protection agency, ethical committee?) Local representatives: local coordination and follow-up. Patient notes review. Additional secretarial assistance, paid or unpaid, is permitted.

Definitions

ESRD

A patient has ESRD if any of the following:

1. He receives a transplant
2. The doctor "believes" that he has ESRD at first dialysis
3. He has received >90 days dialysis
4. If the doctor is in doubt whether the patient has acute or chronic renal failure, the patient is registered as soon as there is no doubt that the patient has ESRD For 3 & 4, registration is performed retrospectively from the first dialysis day.

Planned dialysis

The patient's first dialysis is planned if:

1. His first hemodialysis uses an AV fistula
2. His first hemodialysis uses a permanent catheter as the patient's permanent access
3. His first peritoneal dialysis is >6 days after catheter placement.

The patient's first dialysis is unplanned if:

1. His first hemodialysis uses a temporary catheter
2. His first hemodialysis uses a permanent catheter as the patient's temporary access (i.e. a later AV fistula is planned.
3. His first peritoneal dialysis is <7 days after catheter placement.

Renal Diagnoses

1. Shrunken Kidneys of unknown cause
2. Glomerulonephritis
3. Chronic interstitial nephropathy, chronic pyelonephritis and postrenal uremia
4. Polycystic kidney disease
5. Hypertensive/atherosclerotic renal disease
6. Diabetic Nephropathy
7. Other

Causes of unplanned dialysis

1. Late referral
2. Acute uremia
3. Acute progression of chronic uremia
4. Doubt about reversibility
5. Clinical indication despite acceptable biochemistry
6. Fistula problems
7. Delayed planning (Controversial. I recommend dialysis planning at the latest when eGFR <15 ml/minute. Please use your own definition).
8. Patient non-compliance
9. Patient refused dialysis, but later changed his/her mind

Causes of PD modality

1. Patient choice
2. Cardiac insufficiency
3. HD not possible

Causes of HD Modality

1. Patient Choice
2. Physically incapable of peritoneal dialysis (PD)
3. Mentally incapable of PD
4. Abdominal problems
5. Wish for Home HD
6. PD not considered

Table 1 Center Questionnaire

1. Author:
2. Centre Name:
3. Centre type: University/Non-academic
4. Approximate population covered:
5. No. new ESRD patients/year
6. How many of these

   1. Preemptive transplant (%)?
   2. PD (%)?
   3. HD (%)?
7. What is the

   1. PD prevalence (no. patients)?
   2. HD prevalence?
8. How many nephrology specialists?
9. Does the department have an official policy concerning preferred initial modality:

   1. No
   2. PD first
   3. Home HD first
   4. Other (what?)
10. Does the department have an official policy concerning when pretransplant investigations should be initiated? If so what? If not, is there unofficial consensus? What?
11. Does the department have an official policy concerning when dialysis modality choice is made? If so what? If not, is there unofficial consensus? What?
12. Does the department have an official policy concerning when AV fistulae/grafts are prescribed? If so what? If not, is there unofficial consensus? What?
13. Does the department have an official policy concerning when peritoneal dialysis catheters are prescribed? If so what? If not, is there unofficial consensus? What?
14. Does the department have an official policy concerning when chronic dialysis is prescribed? If so what? If not, is there unofficial consensus? What?

Table 2. Motivation Questionnaire

You have just prescribed this patient's first dialysis. If you do not believe that the patient's dialysis requirement is chronic, you do not have to fill in this form Put a "1" besides the primary reason for starting dialysis today. Put a "2" besides a (possible) secondary reason for starting dialysis today. Put a "X" besides any other reasons that have been important in influencing your decision to prescribe dialysis today.

Taste disturbances Pulmonary stasis Social (what?) Dyspnea Practical (what?) (e.g. catheter protection) Hypertension Pericarditis Oedema Biochemical Cardiac symptoms High Plasma-Creatinine Fatigue High Urea Anorexia Low glomerular filtration rate (GFR) Nausea/vomiting High Potassium Cachexia/weight loss Acidosis Itching Low calcium Insomnia High Calcium Depression High Phosphate Diarrhea Falling GFR Other (what?)

Table 4. Physician Questionnaire What is your age? What is your sex? Are you a nephrology specialist? How many years have you been a doctor? How many years have you been a nephrology specialist?

ELIGIBILITY:
Inclusion Criteria:

* All patients starting maintenance dialysis therapies at the participating centers

Exclusion Criteria:

* Africans

Ages: 1 Month to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Chronic Kidney Disease Stage 5 WHO start dialysis therapy for ESRD
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who start planned dialysis initiation as defined by the protocol | 1 year
  Planned dialysis
  The patient's first dialysis is planned if:
  1. His first hemodialysis uses an AV fistula
  2. His first hemodialysis uses a permanent catheter as the patient's permanent access
  3. His first peritoneal dialysis is >6 days after catheter placement.
  The patient's first dialysis is unplanned if:
  1. His first hemodialysis uses a temporary catheter
  2. His first hemodialysis uses a permanent catheter as the patient's temporary access (i.e. a later AV fistula is planned.
  3. His first peritoneal dialysis is <7 days after catheter placement.

SECONDARY OUTCOMES:
Death | 1 year
  Time to patient death
Choice of dialysis modality | 1 year
  Centre HD, Home HD, CAPD or APD
Choice of dialysis access | 1 year
  AVF, AVG, Temporary CVC, Tunneled CVC, or PD catheter

CONTACTS AND LOCATIONS:
Overall Officials: James G Heaf, MD DMSc, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No